CLINICAL TRIAL: NCT06745895
Title: Multilevel Action Toward Colorectal Cancer and Hepatitis C Education and Screening (MATCHES)
Brief Title: Multilevel Action Toward Colorectal Cancer and Hepatitis C Education and Screening
Acronym: MATCHES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Florida Biomedical Research Program - Bankhead Coley (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: MCC-23232
Record Dates: First submitted 2024-12-17; First posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Colorectal Cancer Screening; Hepatitis C Virus
Keywords: Screening; HCV Screening; CRC Screening; Colorectal Cancer (CRC); Hepatitis C Virus (HCV)
MeSH Terms: conditions — Hepatitis C; Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Eligible and enrolled patient participants enrolled in the intervention will receive a theory-informed educational booklet about both Colorectal Cancer (CRC) and Hepatitis C Virus (HCV) screening in English or Spanish, access to free stool-based CRC screening, and access to HCV screening. Implementation outcomes, facilitators, and barriers will be examined.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multilevel Action Toward Colorectal Cancer and Hepatitis C Education and Screening (MATCHES) (Experimental): The MATCHES intervention includes three patient-level intervention strategies that will be rolled out in two waves. Patient-level strategies are: 1) a combined education booklet with information about CRC/CRC screening and HCV infections/liver cancer/HCV screening in English or Spanish, 2) access to free stool-based CRC screening, and 3) access to free HCV antibody testing.
  Interventions: Behavioral: MATCHES

INTERVENTIONS:
Behavioral: MATCHES — Participants will be asked to complete a survey with specific topics including Hepatitis C (HCV) and Colorectal (CRC) knowledge and health beliefs, screening intentions and demographic characteristics.
  Participants will be provided with education intervention materials (for example, a booklet) either in-person or via mail, access to free stool-based CRC screening, and access to free HCV screening.
  Approximately 1-2 weeks after receiving the education materials, participants will be asked to complete a post-intervention survey about the same specific topics (for example, HCV and CRC knowledge, HCV and CRC health beliefs, HCV and CRC screening intentions, healthcare experiences, perceptions of the educational materials) over the phone with a trained study staff.
  Participants with a positive HCV screening and/or CRC screening result will be navigated to follow-up care as needed.

SUMMARY:
This innovative Multilevel Action Toward Colorectal Cancer (CRC) and Hepatitis C Virus (HCV) Education and Screening (MATCHES) intervention aims to promote concurrent HCV and CRC screening among FQHC patients ages 45-75.

DETAILED DESCRIPTION:
While this is a multi-level intervention study, only information related to the patient-level intervention is being reported for the purposes ClinicalTrials.gov.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be receiving care at one of the participating FQHC clinics.
* Participants must be 45-75 years of age.
* Participants must not be up to date with Colorectal Cancer (CRC) screening recommendations such as no colonoscopy in the past 10 years, occult blood test in the past 12 months.
* Participants must never have had Hepatitis C Virus (HCV) antibody screening.
* Participants must be able to read, write, and understand English or Spanish.
* Participants must have no personal history of CRC or current presumptive CRC symptoms such as unresolved rectal bleeding or abdominal pain/bloating.
* Participants must be at average risk for CRC (no hereditary CRC syndromes such as lower gastrointestinal (GI) bleeding, persistent diarrhea, bloating, or lower GI pain, no strong family history of CRC).
* Participants must be asymptomatic for HCV.
* Participants receiving intervention materials must be able and willing to complete surveys and receive the patient level intervention.
* Participants completing qualitative interviews must be willing to complete a remote interview via phone or teleconference software such as ZOOM.
* Participants completing qualitative interviews must be willing to be audio recorded.
* Participants recruited for qualitative interviews only (did not receive MATCHES intervention materials) must have a clinic visit within prior two months.
* All Participants must be able to provide informed consent.

Exclusion Criteria:

* Participants that do not meet all Inclusion Eligibility requirements will be excluded.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Screening Uptake for Hepatitis C Virus (HCV) and Colorectal Cancer (CRC) | Up to 12 Months
  Screening Uptake will be measured by the number of participants who complete both CRC and HCV screening documented via Electronic Health Record (EHR) at 12 months post-intervention.

SECONDARY OUTCOMES:
Screening Completion for Hepatitis C Virus (HCV) | Up to 41 Months
  Screening Completion for HCV will be measured by the number of participants who complete HCV Screening at any time during the Study Period.
Screening Completion for Colorectal Cancer (CRC) | Up to 41 Months
  Screening Completion for CRC will be measured by the number of participants who complete CRC Screening at any time during the Study Period.
Screening Test Results for Hepatitis C (HCV) | Up to 41 Months
  Screening Test Results will be measured as abnormal vs normal
Screening Test Results for Colorectal Cancer (CRC) | Up to 41 Months
  Screening Test Results will be measured as abnormal vs normal
Completion of repeat CRC Screening | Up to 41 Months
  Completion of any repeat CRC Screening will be measured by the number of participants who repeat CRC Screening during the Study interval.

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Christy, PhD, Principal Investigator — Moffitt Cancer Center; Clement K. Gwede, PhD, MPH, RN, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trials website — http://www.moffitt.org/clinical-trials-research/clinical-trials/